CLINICAL TRIAL: NCT02198456
Title: Prostanoid Therapy in Severe Pulmonary Arterial Hypertension - Imaging Control Study, 3D Echo, MR and RHC.
Brief Title: Imaging Control Study, 3D Echo, MR and RHC.
Acronym: PARIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Steringer-Mascherbauer (Other)
Responsible Party: Sponsor-Investigator, Regina Steringer-Mascherbauer, OA Dr., Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Other Study IDs: Protocol PARIS3D
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Arterial Hypertension WHO Group I
Keywords: pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3D echocardiography

SUMMARY:
The aim of the study is to intensify the follow up of patients with pulmonary arterial hypertension via modern imaging guided methods in due consideration of the possibilities of three-dimensional echocardiography in order to optimize their specific therapy.

The hypothesis is that the increased use of modern imaging guided tools is essential for the follow up.

DETAILED DESCRIPTION:
It is not possible to perform a magnetic resonance imaging in all patients and as a result echocardiography is not only done at screening but also during the follow up. The imaging technologies made a great progress in the last few years and enable a better assessment of the haemodynamic parameters in our days.

ELIGIBILITY:
Inclusion Criteria:

* age >17
* pulmonary arterial hypertension WHO group I who are going to start a therapy with prostanoid
* written informed consent
* Prostanoid naive
* no change of the pulmonary arterial hypertension therapy within 3 weeks of inclusion into the study

Exclusion Criteria:

* pregnancy and lactation period
* Women of childbearing potential who do not use an effective and secure method for birth control
* severe chronic kidney insufficiency (glomerular filtration rate <30), which will remain for more than 3 months
* liver insufficiency Child C
* life expectancy shorter than the course of the study (for example because of a malignant disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary arterial hypertension WHO group I
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
right ventricular ejection fracture | month 12 (+/- 7 days)
  right-sided heart catheterization

SECONDARY OUTCOMES:
right atrial pressure | 12 month (+/- 7 days)
  right-sided heart catheterization
cardiac index (CI)/cardiac output (CO) | 12 months (+/- 7 Days)
  right-sided heart catheterization
pulmonary vascular resistance | 12 months (+/- 7 days)
  right-sided heart catheterization
mean pulmonary capillary wedge pressure | 12 month (+/-7 days)
  right-sided heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steringer-Mascherbauer, MD, Principal Investigator — Krankenhaus der Elisabethinen Linz GmbH
Locations (1):
- Krankenhaus der Elisabethinen Linz GmbH, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided